CLINICAL TRIAL: NCT02928640
Title: Prospective, Multi-Center Study of the ClariCore Optical Biopsy System in Patients Undergoing TRUS-Guided Prostrate Biopsy With or Without MR Fusion For Prostrate Tissue Classification Algorithm Development
Brief Title: ClariCore Optical Biopsy System Used in TRUS (Trans-Rectal Ultrasound)-Guided Prostrate Biopsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Precision Biopsy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIP-1010
Record Dates: First submitted 2016-10-04; First posted 2016-10-10 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Cellular Diagnosis, Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ClariCore System (Experimental): ClairCore System study designed for data collection to build the prostrate tissue classification algorithm.
  Interventions: Device: ClariCore System

INTERVENTIONS:
Device: ClariCore System — Data collection to build the prostrate tissue classification algorithm.
  Other Names: ClariCore Optical Biopsy System

SUMMARY:
The purpose of the study is to collect information on prostrate biopsy tissue for use in developing a method determining the difference in normal and cancerous prostrate tissue using the ClariCore System.

DETAILED DESCRIPTION:
The purpose of this study is to collect information on prostrate tissue biopsies using the ClariCore System. The ClariCore system is designed to improve how the tissue samples are being collected from the prostrate by using light sensors (fiber optics) that can see changes in the tissue. Researchers will study the data collected from the light sensor (optical readings) to develop a method (like a mathematical equation) that can be used to tell the difference between normal and cancerous prostrate tissue during the biopsy. What the researchers are hoping to learn from this study is if a light guided biopsy procedure can improve the accuracy of prostrate biopsy sampling.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for TRUS-guided prostrate biopsy with or without MR TRUS Fusion determined based on standard of care requirements
* Prostrate volume ≥ 20cc and height at least 22mm (at the area(s) to be biopsied) as verified by ultrasound or prostrate MRI
* Patient, or authorized representative signs a written Informed Consent form to participate in the study, prior to any study mandated determinations or procedure

Exclusion Criteria:

* Contraindications to TRUS prostrate biopsy

  * Acute painful perianal disorder
  * Surgical absence of a rectum or the presence of a rectal fistula
* Patients with contraindications to MRI (e.g., pacemaker, claustrophobia, etc.) (MR/TRUS only)

  ---Patients with renal dysfunction are excluded due to their inability to undergo contrast enhanced MRI
* Previous prostrate surgeries
* Prior pelvic irradiation
* Active inflammatory bowel disease within the last 6 months
* Any condition, or history of illness or surgery that, in the opinion of the Investigator, might confound the results of the study or pose additional risks to the patient (e.g., significant cardiovascular conditions or allergies)
* Patient has systemic infection or evidence of any surgical site infection (superficial or organ space), including active urinary tract infection
* Bladder cancer (current or prior)
* Symptomatic acute prostatitis
* Actively taking blood thinning agents (with the exception of low dose aspirin [81 mg] Plavix, Coumadin, etc.) or severe comorbidity prohibiting halting of anticoagulation therapies or history of bleeding disorder (e.g., coagulopathy
* Any malignancy other than non-melanoma cell skin cancer, unless no evidence of disease for a minimum of 5 years
* Hormone therapy for locally advanced disease (except patients on 5-alpha reductase inhibitors to reduce the size of the prostrate)
* Neo-adjuvant hormonal therapy
* Salvage radical prostatectomy, i.e., patients having surgery due to failure of previous therapy (radiation, brachytherapy, cryotherapy, etc.)
* Patient has a compromised immune system or autoimmune disease (WBC < 4000 or > 20,000)
* Patient is not likely to comply with the follow-up evaluation schedule
* Patient is participating in a clinical trial of another investigational drug or device
* Patient is mentally incompetent or a prisoner

Min Age: 22 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-09; Primary Completion 2020-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness | Ath the time of procedure
  Correlate histopathology of tissue biopsy core samples with corresponding spectral data obtained in vivo for algorithm training at time of procedure.

SECONDARY OUTCOMES:
Assessment of Pain | Up to 30 days post-procedure
  Pain shall be reported based on the patient-reported level of pain during the ClariCore System procedure and at 7 and 30 days post-procedure as measured on a 10 point numerical rating scale (NRS).
Incidence and frequency of adverse events | Up to 30 days post-procedure
  The secondary safety endpoint is the incidence and frequency of all Adverse Event's (both related and unrelated to the ClariCore System) reported during the study.

OTHER OUTCOMES:
Technical Success | Until clinical study closure, at time of 30 day follow up
  Ability to obtain optical spectra: defined as the ability to obtain the optical spectra of underlying tissue at each target site and record and store the data on the software and obtain viable biopsy sample from the underlying tissue where the optical spectra data were collected: defined as a sample that the pathologist can use to classify the specific tissue.
Clinical Success | Until clinical study closure, at time of 30 day follow up
  Clinical success is defined at the biopsy core level as the device's ability to obtain a technically successful core and an accurate correlation with optical spectra for the purpose of the tissue classification development.
Negative Predictive Value | Until clinical trial closure, at time of 30 days follow up
  The negative predictive value (NPV) will be estimated as a function of prevalence.

CONTACTS AND LOCATIONS:
Overall Officials: Sierra Yearly, Study Director — Sponsor GmbH
Locations (5):
- United States (5):
  - The Urology Center of Colorado, Denver, Colorado
  - Johns Hopkins Brady Urological Institute- The Johns Hopkins Hospital, Baltimore, Maryland
  - Comprehensive Urology, Royal Oak, Michigan
  - Associated Professionals of New York, PLLC, Syracuse, New York
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina

IPD SHARING:
Plan to Share IPD: No